CLINICAL TRIAL: NCT06593587
Title: A PHASE 3 STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF RESPIRATORY SYNCYTIAL VIRUS (RSV) PREFUSION F SUBUNIT VACCINE IN OLDER ADULTS IN KOREA
Brief Title: A Study to Assess the Safety, Tolerability, and Immunogenicity of RSVpreF in Older Adults in Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3671053; NCT06593587 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Virus
Keywords: Respiratory tract infection; RSV; Respiratory Syncytial Virus; Vaccine; Older adults
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blinded.
  The participant, study coordinator, and all site staff will be blinded.
  The majority of sponsor staff will be blinded to study intervention allocation. All laboratory testing personnel performing serological assays or diagnostic assays will remain blinded to the study intervention assigned/received throughout the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- RSVpreF (Experimental)
  Interventions: Biological: RSVpreF Vaccine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RSVpreF Vaccine — RSV Vaccine 120 mcg
  Arms: RSVpreF
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to quantify the immune response in older Korean adults after a RSVpreF vaccination. It will also learn about the safety and tolerability of RSVpreF vaccination. The main questions it aims to answer are:

What local reactions and systemic events do participants have after a RSVpreF vaccination? What medical problems do participants have after a RSVpreF vaccination? Researchers will compare RSVpreF to a placebo (a look-alike substance that contains no RSVpreF) to see if RSVpreF is safe and well tolerated. It will also examine the change in antibody levels (immune responses) before and after vaccination.

Participants will:

Receive the RSVpreF vaccination or a placebo injection once at Visit 1. Visit the clinic a month later for a checkup and tests. Receive a phone call 1 week after vaccination, and 2 months after vaccination, for health checks.

Keep a diary of their symptoms for 7 days after vaccination.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blinded, placebo-controlled, multicenter trial to describe the safety, tolerability, and immunogenicity of bivalent RSVpreF in adults 60 years of age and older in Korea.

The study duration is approximately 2 months. 4 study visits are required and are comprised of 2 scheduled clinic visits and 2 scheduled telephone calls.

Approximately 360 study-eligible participants will be randomized to receive either the 120-µg dose of RSVpreF or placebo in a 2:1 ratio.

After screening and confirmation of eligibility, a prevaccination blood sample will be collected for immunogenicity assessments and a single dose of study intervention (RSVpreF or placebo) will be administered.

Participants will report daily reactogenicity data using an electronic device for 7-days or until resolution.

Participants will return approximately 1 month later for a follow-up blood draw for immunogenicity assessments and collection of safety information.

A telephone follow-up visit will be conducted approximately 1 week after vaccination to review reactogenicity and approximately 2 months after vaccination to collect safety information.

For all participants, adverse events (AEs) will be collected from informed consent through 1 month following study intervention administration. Serious adverse events (SAEs) newly diagnosed chronic medical conditions (NDCMCs), and adverse events of special interest (AESIs) will be collected from informed consent throughout study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 60 years of age or older at Visit 1

   * Male participants able to father children must agree to use a highly effective method of contraception from the time of informed consent through at least 28 days after study intervention administration
   * Female participants must not be of childbearing potential
2. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

   Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.
3. Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, frequent symptom assessment by mobile device application (e-diary), and other study procedures.
4. Participants who are ambulatory and live in the community, or in assisted-living or long-term care residential facilities that provide minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living (ADL).
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and the protocol.

Exclusion Criteria:

1. A confirmed diagnosis of RSV infection ≤180 days before study intervention administration.
2. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular (IM) injection.
3. Prior history of any subtype of Guillain-Barré syndrome (GBS) of any etiology.
4. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s) or any related vaccine.
5. Serious chronic disorder, including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
6. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
7. Any medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality, that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Individuals who receive chronic systemic treatment with immunosuppressive therapy (other than systemic corticosteroids meeting the criteria noted below), including cytotoxic agents, immunosuppressive monoclonal antibodies, or radiotherapy, eg, for cancer or an autoimmune disease, from 60 days before study intervention administration or planned receipt throughout the study.

   * Receipt of systemic corticosteroids (≥20 mg/day of prednisone or equivalent) for

     ≥14 days from 28 days before study intervention.
   * Inhaled/nebulized, intra articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
9. Receipt of blood/plasma products or immunoglobulin within 60 days before study intervention administration.
10. Previous vaccination with any licensed or investigational RSV vaccine, or planned receipt throughout the study.
11. Previous administration with an investigational product (drug or vaccine) within 6 months prior to study intervention administration. Participation in other studies involving an investigational product (drug or vaccine) at any time during participation in this study.
12. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

    -

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- South Korea (16):
  - Inha University Hospital, Incheon, Incheon-gwangyeoksi [incheon]
  - Jeonbuk National University Hospital, Jeonju, Jeonrabugdo
  - Chonnam National University Hospital, Gwangju, Kwangju-kwangyǒkshi
  - Korea University Ansan Hospital, Ansan-si, Kyǒnggi-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Kyǒnggi-do
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Dong-A University Hospital, Busan, Pusan-kwangyǒkshi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Hallym University Kangdong Sacred Heart Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Hallym University Kangnam Sacred Heart Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Hospital, Daegu, Taegu-kwangyǒkshi

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 16 sites in the Republic of Korea.
Pre-assignment Details: A total of 384 participants were screened, out of which 6 were screen failures and 378 participants were randomized 2:1 to receive respiratory syncytial virus stabilized prefusion F subunit vaccine (RSVpreF) or placebo.
Groups:
- RSVpreF 120 mcg: Participants were randomized to receive a single dose of RSVpreF 120 microgram (mcg) intramuscularly on Day 1.
- Placebo: Participants were randomized to receive a single dose of placebo intramuscularly on Day 1.
Period: Overall Study
Arm/Group | RSVpreF 120 mcg | Placebo
Started | 252 | 126
Vaccinated | 251 | 126
Completed | 250 | 126
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Randomized, not vaccinated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all screened participants who received the study intervention in the study.
Groups:
- RSVpreF 120 mcg: Participants were administered a single dose of RSVpreF 120 mcg on Day 1 via IM injection.
- Placebo: Participants were administered a single dose of placebo on Day 1 via IM injection.
- Total: Total of all reporting groups
Arm/Group | RSVpreF 120 mcg | Placebo | Total
Number analyzed (Participants) | 251 | 126 | 377
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (5.18) | 67.3 (5.19) | 67.3 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 76 | 244
  Male | 83 | 50 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 251 | 126 | 377
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic/non-Latino | 251 | 126 | 377

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination
Description: Local reactions included redness, swelling and pain at injection site. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit=0.5 centimeter (cm). Redness and swelling were graded as mild: > 2.0 cm to 5.0 cm, moderate: > 5.0 cm to 10.0 cm, severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with activity, moderate: interfered with activity, severe: prevented daily activity. Any local reaction: any redness, any swelling, or pain at the injection site of at least mild severity. Exact 2-sided 95% confidence interval (CI) was based on the Clopper and Pearson method.
Time Frame: From Day 1 to Day 7 after vaccination
Population: Safety population included all screened participants who received the study intervention in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg | Placebo
Number analyzed (Participants) | 251 | 126
Percentage of participants
  Pain at injection site: any | 12.4 [8.5 to 17.1] | 3.2 [0.9 to 7.9]
  Pain at injection site: mild | 11.6 [7.9 to 16.2] | 2.4 [0.5 to 6.8]
  Pain at injection site: moderate | 0.8 [0.1 to 2.8] | 0.8 [0.0 to 4.3]
  Pain at injection site: severe | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Redness: any | 2.8 [1.1 to 5.7] | 0.8 [0.0 to 4.3]
  Redness: mild | 1.6 [0.4 to 4.0] | 0.8 [0.0 to 4.3]
  Redness: moderate | 0.8 [0.1 to 2.8] | 0 [0.0 to 2.9]
  Redness: severe | 0.4 [0.0 to 2.2] | 0 [0.0 to 2.9]
  Swelling: any | 1.6 [0.4 to 4.0] | 0.8 [0.0 to 4.3]
  Swelling: mild | 1.2 [0.2 to 3.5] | 0.8 [0.0 to 4.3]
  Swelling: moderate | 0.4 [0.0 to 2.2] | 0 [0.0 to 2.9]
  Swelling: severe | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Any local reaction: any | 14.7 [10.6 to 19.7] | 3.2 [0.9 to 7.9]
  Any local reaction: mild | 12.4 [8.5 to 17.1] | 2.4 [0.5 to 6.8]
  Any local reaction: moderate | 2.0 [0.6 to 4.6] | 0.8 [0.0 to 4.3]
  Any local reaction: severe | 0.4 [0.0 to 2.2] | 0 [0.0 to 2.9]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events included fever, fatigue, headache, vomiting, nausea, diarrhea, muscle pain and joint pain. Fever defined as oral temperature >=38.0 degrees Celsius (deg C) and categorized as mild: >=38.0 to 38.4 deg C, moderate: >38.4 to 38.9 deg C, severe: >38.9 to 40.0 deg C, and Grade 4: >40.0 deg C. Vomiting categorized as mild: 1-2 times in 24 hours (h); moderate: >2 times in 24h; severe: required intravenous (IV) hydration. Diarrhea categorized as mild: 2-3 loose stools in 24h; moderate: 4-5 loose stools in 24h; severe: 6 or more loose stools in 24h. Headache, fatigue, nausea, muscle pain and joint pain were categorized as mild: didn't interfere with activity; moderate: some interference with activity; severe: prevented daily routine activity. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: From Day 1 to Day 7 after vaccination
Population: Safety population included all screened participants who received the study intervention in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg | Placebo
Number analyzed (Participants) | 251 | 126
Percentage of participants
  Fever: >=38.0°C | 0.4 [0.0 to 2.2] | 1.6 [0.2 to 5.6]
  Fever: >=38.0°C to 38.4°C | 0 [0.0 to 1.5] | 1.6 [0.2 to 5.6]
  Fever: >38.4°C to 38.9°C | 0.4 [0.0 to 2.2] | 0 [0.0 to 2.9]
  Fever: >38.9°C to 40.0°C | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Fever: >40.0°C | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Fatigue: any | 23.1 [18.0 to 28.8] | 26.2 [18.8 to 34.8]
  Fatigue: mild | 17.9 [13.4 to 23.2] | 15.9 [10.0 to 23.4]
  Fatigue: moderate | 5.2 [2.8 to 8.7] | 10.3 [5.6 to 17.0]
  Fatigue: severe | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Headache: any | 12.7 [8.9 to 17.5] | 11.1 [6.2 to 17.9]
  Headache: mild | 11.6 [7.9 to 16.2] | 8.7 [4.4 to 15.1]
  Headache: moderate | 1.2 [0.2 to 3.5] | 2.4 [0.5 to 6.8]
  Headache: severe | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Muscle pain: any | 15.5 [11.3 to 20.6] | 9.5 [5.0 to 16.0]
  Muscle pain: mild | 12.0 [8.2 to 16.6] | 5.6 [2.3 to 11.1]
  Muscle pain: moderate | 3.6 [1.7 to 6.7] | 4.0 [1.3 to 9.0]
  Muscle pain: severe | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Joint pain: any | 9.2 [5.9 to 13.4] | 7.9 [3.9 to 14.1]
  Joint pain: mild | 6.0 [3.4 to 9.7] | 4.0 [1.3 to 9.0]
  Joint pain: moderate | 3.2 [1.4 to 6.2] | 4.0 [1.3 to 9.0]
  Joint pain: severe | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Nausea: any | 3.6 [1.7 to 6.7] | 6.3 [2.8 to 12.1]
  Nausea: mild | 3.6 [1.7 to 6.7] | 4.0 [1.3 to 9.0]
  Nausea: moderate | 0 [0.0 to 15] | 2.4 [0.5 to 6.8]
  Nausea: severe | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Vomiting: any | 0 [0.0 to 1.5] | 0.8 [0.0 to 4.3]
  Vomiting: mild | 0 [0.0 to 1.5] | 0.8 [0.0 to 4.3]
  Vomiting: moderate | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Vomiting: severe | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Diarrhea: any | 4.8 [2.5 to 8.2] | 4.0 [1.3 to 9.0]
  Diarrhea: mild | 4.8 [2.5 to 8.2] | 4.0 [1.3 to 9.0]
  Diarrhea: moderate | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]
  Diarrhea: severe | 0 [0.0 to 1.5] | 0 [0.0 to 2.9]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Vaccination Through 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From vaccination on Day 1 up to 1 month after vaccination
Population: Safety population included all screened participants who received the study intervention in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg | Placebo
Number analyzed (Participants) | 251 | 126
Percentage of participants | 3.6 [1.7 to 6.7] | 0.8 [0.0 to 4.3]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Vaccination Throughout the Study
Description: An SAE was defined as an AE that, at any dose met one of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or nonpathogenic; other significant medical events as judged by investigator. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: From vaccination on Day 1 up to 2 months after vaccination
Population: Safety population included all screened participants who received the study intervention in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg | Placebo
Number analyzed (Participants) | 251 | 126
Percentage of participants | 0.8 [0.1 to 2.8] | 0.8 [0.0 to 4.3]

5. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) From Vaccination Throughout the Study
Description: A NDCMC was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects. Newly diagnosed chronic medical condition did not include illnesses considered to be temporary conditions. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: From vaccination on Day 1 up to 2 months after vaccination
Population: Safety population included all screened participants who received the study intervention in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg | Placebo
Number analyzed (Participants) | 251 | 126
Percentage of participants | 1.2 [0.2 to 3.5] | 0 [0.0 to 2.9]

6. Primary Outcome: Geometric Mean Titer (GMT) of Neutralizing Titers (NTs) for RSV A and RSV B Before Vaccination
Description: GMTs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the lower limit of quantification (LLOQ) were set to 0.5*LLOQ for analysis.
Time Frame: Before Vaccination
Population: Evaluable immunogenicity population: all participants who were eligible and received the study intervention to which they were randomized, had 1-month postvaccination blood collection visit within 27 to 42 days after vaccination, had at least 1 valid and determinate assay result 1 month after vaccination and had no major protocol violations from vaccination through the 1-month postvaccination blood draw. Here "Number Analyzed" refers to number of participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSVpreF 120 mcg | Placebo
Number analyzed (Participants) | 249 | 126
Titer
  RSV A: number analyzed (Participants) | 248 | 126
  RSV A | 1472 [1326 to 1636] | 1617 [1402 to 1866]
  RSV B | 1957 [1766 to 2168] | 1865 [1601 to 2174]

7. Primary Outcome: Geometric Mean Titer (GMT) of Neutralizing Titers (NTs) for RSV A and RSV B at 1 Month After Vaccination
Description: GMTs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ for analysis.
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSVpreF 120 mcg | Placebo
Number analyzed (Participants) | 249 | 126
Titer
  RSV A: number analyzed (Participants) | 249 | 125
  RSV A | 14240 [12977 to 15625] | 1397 [1199 to 1628]
  RSV B | 16277 [14623 to 18117] | 1813 [1554 to 2115]

8. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Neutralizing Titers (NTs) for RSV A and RSV B From Before Vaccination to 1 Month After Vaccination
Description: Fold rises was defined as ratios of the results after vaccination to the results before vaccination. GMFRs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution).
Time Frame: From before vaccination to 1 month after vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | RSVpreF 120 mcg | Placebo
Number analyzed (Participants) | 249 | 126
Fold rise
  RSV A: number analyzed (Participants) | 248 | 125
  RSV A | 9.5 [8.51 to 10.67] | 0.9 [0.78 to 0.94]
  RSV B | 8.3 [7.37 to 9.39] | 1.0 [0.89 to 1.06]

9. Secondary Outcome: Seroresponse Rates of Neutralizing Titers (NTs) for RSV A and RSV B at 1 Month After Vaccination
Description: Seroresponse rate was defined as the percentage of participants with a postvaccination NT >=4 times the LLOQ if the baseline titer (before vaccination) was below the LLOQ; or a >=4-fold rise from baseline if the baseline titer was>=LLOQ. 95% CI was based on Clopper-Pearson method.
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg | Placebo
Number analyzed (Participants) | 249 | 126
Percentage of participants
  RSV A: number analyzed (Participants) | 248 | 125
  RSV A | 81.0 [75.6 to 85.7] | 0.8 [0.0 to 4.4]
  RSV B | 75.9 [70.1 to 81.1] | 0.8 [0.0 to 4.3]

ADVERSE EVENTS:
Time Frame: All-cause mortality and SAEs: From vaccination on Day 1 up to 2 months after vaccination. Other AEs (non-systematic assessment): From vaccination on Day 1 up to 1 month after vaccination; Local reactions and systemic events (systematic assessment): From Day 1 to Day 7 after vaccination
Description: Same event may appear as both non-SAE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population included all screened participants who received the study intervention in the study.
Arm/Group | RSVpreF 120 mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/251 | 0/126
Serious Adverse Events (participants affected / at risk) | 2/251 | 1/126
Other Adverse Events (participants affected / at risk) | 100/251 | 43/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSVpreF 120 mcg (N=251) | Placebo (N=126)
Retinal detachment (Eye disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSVpreF 120 mcg (N=251) | Placebo (N=126)
Asthenia (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Fatigue (FATIGUE) (General disorders) | 58 | 33
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 31 | 4
Pyrexia (FEVER) (General disorders) | 1 | 2
Swelling (SWELLING) (General disorders) | 4 | 1
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 12 | 5
Nausea (NAUSEA) (Gastrointestinal disorders) | 9 | 8
Vomiting (VOMITING) (Gastrointestinal disorders) | 0 | 1
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 23 | 10
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 39 | 12
Headache (HEADACHE) (Nervous system disorders) | 32 | 14
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT06593587/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT06593587/SAP_001.pdf